CLINICAL TRIAL: NCT03120728
Title: AFTER: Application for the Etonogestrel/Ethinyl Estradiol Ring--potential for Emergency Contraception
Brief Title: Application for the Etonogestrel/Ethinyl Estradiol Ring
Acronym: AFTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Diana Crabtree Sokol, Principal investigator, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-16-00930
Record Dates: First submitted 2017-03-31; First posted 2017-04-19 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Emergency Contraception; Healthy, Reproductive Age Women
Keywords: Emergency contraception; Contraceptive vaginal ring; NuvaRing; Contraception
MeSH Terms: interventions — etonogestrel; NuvaRing

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 12-14mm leading follicle size (Experimental): Placement of the etonogestrel/ethinyl estradiol contraceptive vaginal ring when leading follicle measures 12-14mm on transvaginal ultrasound.
  Interventions: Drug: Etonogestrel/ethinyl estradiol contraceptive vaginal ring
- 15-17mm leading follicle size (Experimental): Placement of the etonogestrel/ethinyl estradiol contraceptive vaginal ring when leading follicle measures 15-17mm on transvaginal ultrasound.
  Interventions: Drug: Etonogestrel/ethinyl estradiol contraceptive vaginal ring
- 18mm or greater leading follicle size (Experimental): Placement of the etonogestrel/ethinyl estradiol contraceptive vaginal ring when leading follicle measures 18mm or greater on transvaginal ultrasound.
  Interventions: Drug: Etonogestrel/ethinyl estradiol contraceptive vaginal ring

INTERVENTIONS:
Drug: Etonogestrel/ethinyl estradiol contraceptive vaginal ring — Placement of a contraceptive vaginal ring with subsequent assessment of ovulation disruption. Timing of placement depends on leading follicle size, as described in "Arms" section.
  Other Names: NuvaRing; Contraceptive vaginal ring

SUMMARY:
This study is enrolling healthy women ages 18-39yo who are not pregnant or breastfeeding, and are not using hormonal birth control. Initial screening visit will include a blood draw to assess if the participant has recently ovulated. If hormone test indicates ovulation occurred, participant will start the study 8 days after the start of their next menstrual period. On this study visit, vaginal ultrasound will be performed to look the ovaries for follicles. Vaginal ultrasound is then performed approximately every 2 days until the dominant follicle has grown into the size group assigned. When this occurs the participant will place the NuvaRing®, inside the vagina and blood will be drawn for hormone levels. Participant will then return daily the next 5 days (total of 6 daily visits) for vaginal ultrasound and blood draw to assess for signs of ovulation. After the 7th day the ring is in the vagina, the participant will remove the ring from her vagina at home. After removal, there will be twice weekly clinic visits for ultrasound and blood draw until menstrual bleeding occurs. At this point, participation in the study is complete. Participants are compensated for their time.

DETAILED DESCRIPTION:
The study will be comprised of healthy, non-pregnant, non-breastfeeding, reproductive age women with regular, ovulatory cycles who are protected from unintended pregnancy via the concurrent use of non-hormonal methods of contraception. Participants will have a mid-luteal screening visit, which will include: informed consent, history, physical, vitals, and assessment of mid-luteal serum progesterone to confirm ovulatory status. Each participant will be assigned to one of three groups according the size of the leading follicle (12-14mm, 15-17mm, ≥18mm), which will determine the timing of the placement of the ENG/EE CVR. Transvaginal ultrasound (TVUS) will be performed three times per week, starting on day 8 of the menstrual cycle, until the leading follicle is within the assigned group. On that day the CVR will be placed and, including day of placement, there will be 6 daily visits with hormonal assays (progesterone, luteinizing hormone) and TVUS to assess for signs of ovulation. Compliance with CVR placement will be assessed through the measurement of serum ENG. After 7 days, participants will remove the CVR at home. Participants will then have biweekly visits until onset of menses to obtain serum progesterone levels and TVUS to assess for signs of delayed ovulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, women ages 18 to 39yo with BMI <30
* Regular menstrual cycles with duration between 24-35 days
* Completion of screening visit where ovulation will be assessed with blood draw for progesterone level (must be 5ng/mL or greater)
* Not seeking pregnancy during the study period
* Use of a non-hormonal form of contraception, such as: sterilization (tubal ligation, Essure), copper IUD (intrauterine device), barrier methods or abstinence
* Must speak English or Spanish

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Severe pelvic organ prolapse or prolapse to any degree that may prevent retention of the vaginal ring after insertion
* Use of oral contraceptive pills, patches, implants or hormonal intrauterine contraception in the month prior to screening
* Use of depo medroxyprogesterone within 6 months of screening
* Use of medications that interact with contraceptive steroid hormones: anti-epileptic medications, rifampin, rifabutin, fosamprenavir, etc
* Medical condition with safety deemed to be category 3 or 4 when using a combined hormonal contraceptive, as determined by the Center for Disease Control Medical Eligibility Criteria: current or past history of breast cancer, severe decompensated cirrhosis, history of deep vein thrombosis or pulmonary embolus, diabetes with nephropathy/retinopathy/neuropathy or other vascular disease diagnosed more than 20 years ago, current symptomatic gallbladder disease, hypertension, ischemic heart disease, known thrombogenic mutations, hepatocellular adenoma, malignant hepatoma, multiple risk factors for atherosclerotic cardiovascular disease, multiple sclerosis with prolonged immobility, history of peripartum cardiomyopathy, cigarette smoking and ≥35yo, history of complicated solid organ transplant, history of stroke, history of superficial venous thrombosis not associated with catheter, systemic lupus erythematosus with positive antiphospholipid antibodies, valvular heart disease complicated by pulmonary hypertension or atrial fibrillation or bacterial endocarditis, and acute viral hepatitis

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of ovulation suppression or dysfunction in relation to follicle size | The outcome is measured throughout the 6 week study.
  Describe the ability of the contraceptive vaginal ring to cause ovulation suppression or dysfunction when placed in the mid and advanced follicular phase. This will be determined via measurement of steroid hormones and assessment of the leading ovarian follicle for signs of rupture after placement of the contraceptive vaginal ring.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Crabtree Sokol, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Keck Medicine of USC--Downtown LA, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No